CLINICAL TRIAL: NCT03771625
Title: Evaluating Changes of Brain Networks and White Matter Fibers by fMRI and DTI After Treatments in Patients With Germ Cell Tumors in the Basal Ganglia
Brief Title: Evaluating Structural and Functional Changes of Brain by fMRI and DTI in Patients With Intracranial Germ Cell Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-GEMF-1073
Record Dates: First submitted 2018-12-04; First posted 2018-12-11 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2018-12

CONDITIONS: Intracranial Germ Cell Tumor
Keywords: fMRI; DTI; Intracranial Germ cell tumor; Basal ganglia
MeSH Terms: interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single-group studies: All the patients received chemotherapy and radiotherapy.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — whole brain with/without spinal cord
  Other Names: chemotherapy

SUMMARY:
BOLD-fMRI and DTI scans are performed to patients with germ cell tumors in the basal ganglia before and after treatments. The changes of the MRI and muscle strength of patients during treatments are evaluated, and the association between these two are investigated.

DETAILED DESCRIPTION:
Primary intracranial germ cell tumors are a specific entity of brain tumors with a variety of histological types and different degrees of malignancy. Intracranial GCTs make up 11.2% - 15.3% of primary intracranial tumors in Asian children compared with 3.6% in the US. And tumors located at the basal ganglia is much rarer.

The investigators realize that most of patients with tumors at this location are involved with motor disfunction. And after treatments, some patients get relieved dramatically, but some others failed to get similar outcomes. To better understand the mechanism causing this difference of treatment outcomes, the investigators perform BOLD-fMRI and DTI scans to patients with germ cell tumors in the basal ganglia before and after treatments. The changes of the fMRI and muscle strength of patients during treatments are evaluated, and the association between these two are investigated.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥3 years;
2. no history of brain radiotherapy;
3. no other known cause of movement and cognitive impairment;
4. no contraindications to the magnetic resonance imaging (MRI) scan;

Exclusion Criteria:

1. patients can not tolerate MR scan;
2. head motion is greater than 3 mm during functional MRI scanning.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intracranial germ cell tumor located at the basal ganglia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes of brain networks measured by BOLD-fMRI after treatments. | The fMRI scans are performed: (1) before treatments in one week, (2) before radiotherapy in one week, (3) after radiotherapy in one week, (4) one year after radiotherapy.
  The brain networks during treatments are compared by functional connectivity.
Changes of white matter fibers measured by DTI after treatments. | The DTI scans are performed along with the fMRI scans.
  The white matter fibers damaged by tumor are evaluated by FA and MD value.

SECONDARY OUTCOMES:
Changes of muscle strength after treatments. | The muscle strength evaluation are performed at the same day before the fMRI scans.
  The limb muscle strength of patients are evaluated with the Medical Research Council (MRC) scale for muscle strength (grade 0-5).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Background] Liang SY, Yang TF, Chen YW, Liang ML, Chen HH, Chang KP, Shan IK, Chen YS, Wong TT. Neuropsychological functions and quality of life in survived patients with intracranial germ cell tumors after treatment. Neuro Oncol. 2013 Nov;15(11):1543-51. doi: 10.1093/neuonc/not127. Epub 2013 Oct 6. PMID 24101738